CLINICAL TRIAL: NCT01475539
Title: Immunogenicity and Safety of Different Sequential Schedules of Inactivated Poliomyelitis Vaccine (IMOVAX Polio®) Followed by Oral Poliomyelitis Vaccine in Healthy Infants in China Versus Oral Poliomyelitis Vaccine Alone.
Brief Title: Sequential Inactivated Poliomyelitis Vaccine Followed by Oral Poliomyelitis Vaccine Versus Oral Poliomyelitis Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IPV30; U1111-1122-1928 (Other: WHO)
Record Dates: First submitted 2011-11-14; First posted 2011-11-21 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Polio; Poliomyelitis
Keywords: Polio; Poliovirus; Oral poliovirus vaccine; IMOVAX Polio®
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Sequential 1): IPV-OPV-OPV (Experimental): Participants will receive 1 dose of Sanofi Pasteur's injectable Inactivated Poliovirus Vaccine (IPV) followed by 2 doses of a commercially available Oral Poliovirus Vaccine (OPV)
  Interventions: Biological: Injectable inactivated types 1, 2 and 3 poliovirus + Live oral Polio
- Group B (Sequential 2): IPV-IPV-OPV (Experimental): Participants will receive 2 doses of Sanofi Pasteur's injectable Inactivated Poliovirus Vaccine (IPV) followed by 1 dose of a commercially available Oral Poliovirus Vaccine (OPV)
  Interventions: Biological: Injectable inactivated types 1, 2 and 3 poliovirus + Live oral Polio
- Group C (Reference): OPV-OPV-OPV (Experimental): Participants will receive 3 doses of a commercially available Oral Poliovirus Vaccine (OPV)
  Interventions: Biological: Live oral poliovirus type 1, 2 and 3

INTERVENTIONS:
Biological: Injectable inactivated types 1, 2 and 3 poliovirus + Live oral Polio — 0.5 mL, Intramuscular + 1g dragee candy oral dose
  Other Names: IMOVAX Polio®
  Arms: Group A (Sequential 1): IPV-OPV-OPV
Biological: Injectable inactivated types 1, 2 and 3 poliovirus + Live oral Polio — 0.5 mL, Intramuscular + 1g dragee candy oral dose
  Other Names: IMOVAX Polio®
  Arms: Group B (Sequential 2): IPV-IPV-OPV
Biological: Live oral poliovirus type 1, 2 and 3 — 1g dragee candy, oral
  Arms: Group C (Reference): OPV-OPV-OPV

SUMMARY:
The purpose of this study is to generate data to support the registration extension of IMOVAX Polio to be used in a sequential vaccination.

Primary objective:

* To demonstrate the non-inferiority of Inactivated Poliomyelitis Vaccine (IPV)-(Oral Poliomyelitis Vaccine) (OPV)-OPV (Sequential 1) and IPV-IPV-OPV (sequential 2) poliovirus vaccine administrations versus OPV-OPV-OPV (Reference) in terms of seroprotection rate 28 to 42 days after the third dose of the primary vaccination series.

Secondary objectives:

* To evaluate the safety profile of the investigational vaccines after each administration in each group.
* To describe the humoral immune response to poliovirus serotypes (types 1, 2 and 3) before the first dose and 28 to 42 days after the third primary series dose of vaccine in each group.
* To describe the persistence of antibodies against poliovirus serotypes (types 1, 2 and 3) after the third primary series dose administration, at 18 months of age in each group.

DETAILED DESCRIPTION:
Study participants will be randomized to receive either 3 doses of a commercially available Oral Poliovirus Vaccine (OPV), or 1 dose of Sanofi Pasteur's injectable Inactivated Poliovirus Vaccine IMOVAX Polio (IPV) followed by 2 doses of OPV, or 2 doses of IPV followed by 1 dose of OPV.

These vaccines will be administered at 2, 3 and 4 months of age as primary vaccination for the prevention of poliomyelitis. Participants will be followed up through their 18th- to 19th-month birthday.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥2 months and less than 3 months on the day of first study vaccine administration
* Born at full term of pregnancy (≥37 weeks) and with a birth weight ≥2.5 kg
* Informed consent form has been signed and dated by the parent or other legally acceptable representative
* Subject and parent/legally acceptable representative are able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt or planned receipt of any vaccine in the 4 weeks preceding or following any trial vaccination (except Diphtheria, Tetanus, acellular Pertussis vaccine [DTaP], Haemophilus Influenzae Type b [Hib] vaccine, bacille Calmette-Guerin vaccine [BCG] and Hepatitis B given at least 7 days before and after study vaccination)Previous vaccination against poliomyelitis with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products since birth
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy since birth; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks since birth)
* Congenital or acquired immunodeficiency in close contacts to the subjects
* History of poliomyelitis infection (confirmed either clinically, serologically or microbiologically)
* At high risk for human immunodeficiency virus (HIV) infection during the trial
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Laboratory-confirmed or otherwise known thrombocytopenia, contraindicating intramuscular vaccination
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (axillary temperature ≥37.1°C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study
* Any other contraindication as listed in the study vaccines' leaflets.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 456 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Neutralizing antibody titers ≥8 (1/dil) against each of the 3 poliovirus serotypes (types 1, 2 and 3) after the 3 dose primary vaccination series. | 1 month post-dose 3 (primary vaccination series)
  Antibodies to the vaccine antigens will be determined by a microneutralization assay.

SECONDARY OUTCOMES:
Number and percentage of participants reporting solicited injection site and systemic reaction, and serious adverse events after each vaccination with Polio virus vaccine. | Day 0 up to 17 months post-vaccination
  Solicited injection site: Tenderness, Redness, and Swelling. Solicited Systemic reaction: Fever (Temperature), Vomiting, Abnormal crying, Drowsiness, Loss of Appetite, and Irritability.
Geometric mean titers and anti poliovirus 1,2 and 3 individual antibody titers | Day 0 and up to 16 months post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur China
Locations (1):
- Nanning, Guangxi, China

REFERENCES:
- [Derived] Li RC, Li CG, Wang HB, Luo HM, Li YP, Wang JF, Ying ZF, Yu WZ, Shu JD, Wen N, Vidor E. Immunogenicity of Two Different Sequential Schedules of Inactivated Polio Vaccine Followed by Oral Polio Vaccine Versus Oral Polio Vaccine Alone in Healthy Infants in China. J Pediatric Infect Dis Soc. 2016 Sep;5(3):287-96. doi: 10.1093/jpids/piv017. Epub 2015 Apr 16. PMID 26407255
- See also: Related Info — http://www.sanofipasteur.com